CLINICAL TRIAL: NCT02092506
Title: A Randomized Controlled Trial of Triple Therapy Versus Sequential Therapy Versus Concomitant Therapy as First Line Treatment for Helicobacter Pylori Infection
Brief Title: RCT: Triple vs Sequential vs Concomitant Therapy H Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/389/E
Record Dates: First submitted 2014-02-20; First posted 2014-03-20 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)
Keywords: H pylori; therapy
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- triple therapy (Active Comparator): 10 day triple therapy (PPI, amoxicillin 1g, clarithromycin 500mg twice daily)
  Interventions: Drug: 10 day triple therapy
- Concomitant therapy (Active Comparator): 10-day concomitant therapy (PPI, amoxicillin 1g, clarithromycin 500mg, metronidazole 400mg twice daily).
  Interventions: Drug: 10 day sequential therapy
- sequential therapy (Active Comparator): 10-day sequential therapy (PPI and amoxicillin 1 g twice daily x 5 days followed by PPI, clarithromycin 500mg, metronidazole 400mg twice daily x 5days)
  Interventions: Drug: 10 day concomitant therapy

INTERVENTIONS:
Drug: 10 day triple therapy — 10 day triple therapy
  Other Names: Proton pump inhibitors bd; Amoxicillin 1 g bd; Clarithromycin 500mg bd
  Arms: triple therapy
Drug: 10 day sequential therapy — 10 day sequential therapy
  Other Names: Proton pump inhibitors bd; Amoxicillin 1g twice daily for 5 days; followed by clarithromycin 500mg bd for 5 days; Metronidazole 400mg bd for 5 days
  Arms: Concomitant therapy
Drug: 10 day concomitant therapy — 10 day concomitant therapy
  Other Names: Proton pump inhibitors bd; Amoxicillin 1 g bd; Clarithromycin 500 mg bd; Metronidazole 400 mg bd
  Arms: sequential therapy

SUMMARY:
Triple therapy (TT) comprising proton pump inhibitor (PPI), amoxicillin 1g and clarithromycin 500mg twice daily has long been considered one of the standard treatment for H. pylori infection as initial studies demonstrated success rates of > 90% on per protocol analysis (PP) and > 80% on intention to treat (ITT) analysis. However increasing bacterial resistance, especially to clarithromycin, has been reported and there are concerns that the efficacy of TT has decreased. Sequential therapy (ST) is an alternative first line therapy that consists of 5 days of treatment with a PPI and amoxicillin followed by 5-day treatment with the PPI and clarithromycin and metronidazole. The rationale for this approach is that amoxicillin may weaken the bacterial cell wall in the initial phase of treatment, and prevent the development of drug efflux channels that inhibit clarithromycin from binding to ribosomes and thus help to improve the efficacy of clarithromycin in the second phase of treatment. A recent meta-analysis based on mainly European studies showed that the success rate of ST compared to TT was 92.8 - 96% vs. 76.2 - 78.8%. Concomitant therapy (CT) is another alternative first line treatment that consists of 10 days of PPI, amoxicillin, clarithromycin and metronidazole. The rationale for using CT as a first line treatment option is to address the possibility of clarithromycin resistance which is increasingly encountered in clinical practice. Currently there are no randomized controlled studies that compared TT with ST in Singapore, although both regimens are being used in routine clinical practice. The hypothesis is that ST is superior to TT as first line treatment for H. pylori infection.

The study aim to compare 10-day TT versus 10-day ST versus 10-day CT as first line treatment for H. pylori infection in Singapore.

DETAILED DESCRIPTION:
Background Helicobacter pylori is a common infection in Singapore with an overall seroprevalence rate of 31%. The prevalence rate increases with age and exceeds 70% among those more than 65 years of age (1). H pylori is a major pathogen and is associated with development of peptic ulcer disease and gastric malignancies and successful H. pylori eradication has been shown to be important for both primary and secondary prevention of these diseases (2). Triple therapy (TT) comprising proton pump inhibitor (PPI), amoxicillin 1g and clarithromycin 500mg twice daily has long been considered one of the standard treatment for H. pylori infection (2, 3) as initial studies demonstrated success rates of > 90% on per protocol analysis (PP) and > 80% on intention to treat (ITT) analysis . However increasing bacterial resistance, especially to clarithromycin, has been reported and there are concerns that the efficacy of TT has decreased. Sequential therapy (ST) is an alternative first line therapy that consists of 5 days of treatment with a PPI and amoxicillin followed by 5-day treatment with the PPI and clarithromycin and metronidazole. The rationale for this approach is that amoxicillin may weaken the bacterial cell wall in the initial phase of treatment, and prevent the development of drug efflux channels that inhibit clarithromycin from binding to ribosomes and thus help to improve the efficacy of clarithromycin in the second phase of treatment. A recent meta-analysis based on mainly European studies showed that the success rate of ST compared to TT was 92.8 - 96% vs. 76.2 - 78.8% (4). Concomitant therapy (CT) is another alternative first line treatment that consists of 10 days of PPI, amoxicillin, clarithromycin and metronidazole. The rationale for using CT as a first line treatment option is to address the possibility of clarithromycin resistance which is increasingly encountered in clinical practice (5). Currently there are no randomized controlled studies that compared TT with ST in Singapore, although both regimens are being used in routine clinical practice. The hypothesis is that ST is superior to TT as first line treatment for H. pylori infection.

Aim 10-day triple therapy (TT) [twice daily proton pump inhibitors (PPI), amoxicillin 1 g and clarithromycin 500mg] versus 10-day sequential therapy (ST) [5 day PPI and amoxicillin 1g twice daily followed by 5 days PPI, clarithromycin 500mg and metronidazole 400mg twice daily] versus 10-day concomitant therapy (CT) [twice daily PPI, amoxicillin 1g, clarithromycin 500mg and metronidazole 400mg] as first line treatment for H. pylori infection.

Patients and Methods

Study Design:

Prospective randomized controlled study.

Treatment H. pylori infected patients will be randomized to be treated using either 10 day TT (PPI, amoxicillin 1g, clarithromycin 500mg twice daily) or 10-day ST (PPI and amoxicillin 1 g twice daily x 5 days followed by PPI, clarithromycin 500mg, metronidazole 400mg twice daily x 5days) or 10-day CT (PPI, amoxicillin 1g, clarithromycin 500mg, metronidazole 400mg twice daily). The success of treatment will be defined as either a negative carbon urea breath test (CUBT) or negative histology performed more than 4 weeks after completion of treatment. CUBT or histology will be performed based on the clinical indication as determined by the attending physician. All patients should be off PPI for at least 2 weeks, or histamine 2 receptor antagonists for at least 1 week, prior to assessment of the success of treatment, as per standard practice. The compliance to treatment in terms of percentage of drugs taken will be assessed during clinic review.

Antibiotic susceptibility testing For patients with H. pylori infection diagnosed during endoscopy from a positive rapid urease test kit, the material from the test kit will be used sent for antibiotic susceptibility testing whenever it is technically feasible. This may be of value in guiding the choice of antibiotics for second line salvage treatment should first line treatment fails.

Statistical analysis:

A treatment success rate of 80% is regarded as the minimum acceptable threshold for empiric first line therapy. Data from several countries have suggested that the success rate of triple therapy may be lower than 80%, whereas that for concomitant therapy may exceed 90%. Thus for the study to have 80% power with significance level of 5%, the minimum number of patients to be recruited into each arm will be 138 if the highest success rate is 91% and lowest success rate is 79%. Randomization will be performed in blocks of 15. Categorical data will be analysed using Chi-square or Fisher exact test, while continuous data will be analysed using student's t test. A p value of < 0.05 will be taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients newly diagnosed to have H. pylori infection.

Exclusion Criteria:

* known allergy to any of the treatment drugs
* inability to undergo routine test to confirm success of H. pylori eradication
* previous H. pylori therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
H pylori eradication rate | at least 4 weeks up to 24 weeks after finishing course of antibiotics
  H pylori eradication rate

CONTACTS AND LOCATIONS:
Overall Officials: Tiing Leong Ang, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] 1. Fock KM, Ang TL. Epidemiology of Helicobacter pylori infection and gastric cancer in Asia. J Gastroenterol Hepatol 2010;25:479-86. 2. Fock KM, Talley N, Moayyedi P et al. Asia-Pacific consensus guidelines on gastric cancer prevention. J Gastroenterol Hepatol 2008;23:351-65. 3. Fock KM, Katelaris P, Sugano K, et al. Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol 2009;24:1587-600. 4. Malfertheiner P, Megraud F, O'Morain C et al. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut 2007;56:772-81. 5. Malfertheiner P, Bayerdörffer E, Diete U et al. The GU-MACH study: the effect of 1-week omeprazole triple therapy on Helicobacter pylori infection in patients with gastric ulcer. Aliment. Pharmacol Ther 1999;13:703-12. 6. Zanten SJ, Bradette M, Farley A et al. The DU-MACH study: eradication of Helicobacter pylori and ulcer healing in patients with acute duodenal ulcer using omeprazole based triple therapy. Aliment. Pharmacol Ther 1999;13:289-95. 7. Fock KM, Chelvam P, Lim SG. Triple therapy in the eradication of Helicobacter pylori in patients with duodenal ulcer disease: results of a multicentre study in South-East Asia. South-East Asia Multicenter Study Group. Aliment. Pharmacol. Ther. 2000;14:225-31. 8. Gatta L, Vakil N, Leandro G, Di Mario F, Vaira D. Sequential therapy or triple therapy for Helicobacter pylori infection: systematic review and meta-analysis of randomized controlled trials in adults and children. Am J Gastroenterol 2009;104:3069-79. 9. Rimbara E, Fischbach LA, Graham DY. Optimal therapy for Helicobacter pylori infections. Nat Rev Gastroenterol Hepatol 2011;8:79-88.
- [Derived] Ang TL, Fock KM, Song M, Ang D, Kwek AB, Ong J, Tan J, Teo EK, Dhamodaran S. Ten-day triple therapy versus sequential therapy versus concomitant therapy as first-line treatment for Helicobacter pylori infection. J Gastroenterol Hepatol. 2015 Jul;30(7):1134-9. doi: 10.1111/jgh.12892. PMID 25639278